CLINICAL TRIAL: NCT04107194
Title: Comparison Between Tailored Therapy Guided by a Non-invasive Antibiotic Susceptibility Test and Empiric Treatment for First-line Helicobacter Pylori Eradication in Patients With Dyspepsia: a Randomized Controlled Trial.
Brief Title: Non-invasive Test-guided Tailored Therapy Versus Empiric Treatment for Helicobacter Pylori Infection.
Acronym: THD-HP
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Bari (Other)
Responsible Party: Principal Investigator, Alfredo Di Leo, Professor of University of Bari, University of Bari
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Policlinic Hospital 6, Bari
Record Dates: First submitted 2019-09-25; First posted 2019-09-27 (Actual); Last update posted 2021-01-12 (Actual); Status verified 2021-01

CONDITIONS: Helicobacter Pylori Infection; Antibiotic Resistant Infection; Antibiotic Resistant Strain
MeSH Terms: interventions — Pantoprazole; Amoxicillin; Clarithromycin; Metronidazole; Tetracycline; bismuth tripotassium dicitrate; Rifabutin; Levofloxacin

STUDY DESIGN:
Intervention Model Description: Open-label, multicenter, parallel-arm randomized controlled trial
Who Masked: Outcomes Assessor
Masking Description: Investigators performing urea breath test 30 days after the end of the treatment (assessment of the primary outcome: eradication rate) will not be aware of participants' allocation and received therapy. Moreover, two independent investigators will perform RT-PCR on stool samples and gastric biopsy specimens, blinded to the other test results.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tailored therapy (Experimental): 1. Clarithromycin-sensitive strain (10 day-therapy):
     Pantoprazole 40 mg bid (tablet) Amoxicillin 1000 mg bid (tablet) Clarithromycin 500 mg bid (tablet) Metronidazole 500 mg bid (tablet)
  2. Clarithromycin-resistant and tetracycline-sensitive strain (10 day-therapy):
     Pantoprazole 40 mg bid (tablet) Tetracycline 125 mg + metronidazole 125 mg + bismuth 140 mg in a single tablet (3 tablets qid)
  3. Clarithromycin- and tetracycline-resistant and levofloxacin-sensitive strain (10 day- therapy):
     Pantoprazole 40 mg bid (tablet) Amoxicillin 1000 mg bid (tablet) Levofloxacin 500 mg bid (tablet)
  4. Clarithromycin-, tetracycline- and levofloxacin-resistant strain (10 day-therapy):
  Pantoprazole 40 mg bid (tablet) Amoxicillin 1000 mg bid (tablet) Rifabutin 150 mg bid (tablet)
  Interventions: Drug: Pantoprazole 40mg; Drug: Amoxicillin 1000 MG; Drug: Clarithromycin 500mg; Drug: Metronidazole; Drug: Tetracycline 125 MG; Drug: Bismuth Subcitrate; Drug: Rifabutin 150 MG; Drug: Levofloxacin 500mg
- Empiric therapy (Active Comparator): Either one of the two following 10-day regimens (according to physician's decision):
  1. Pantoprazole 40 mg bid (tablet) Amoxicillin 1000 mg bid (tablet) Clarithromycin 500 mg bid (tablet) Metronidazole 500 mg bid (tablet)
  2. Pantoprazole 40 mg bid (tablet) Tetracycline 125 mg + metronidazole 125 mg + bismuth 140 mg in a single tablet (3 tablets qid)
  Interventions: Drug: Pantoprazole 40mg; Drug: Amoxicillin 1000 MG; Drug: Clarithromycin 500mg; Drug: Metronidazole; Drug: Tetracycline 125 MG; Drug: Bismuth Subcitrate

INTERVENTIONS:
Drug: Pantoprazole 40mg — Proton pump inhibitor
  Other Names: Pantorc
Drug: Amoxicillin 1000 MG — Antibiotic
  Other Names: Zimox
Drug: Clarithromycin 500mg — Antibiotic
  Other Names: Klacid
Drug: Metronidazole — Antibiotic
  Other Names: Flagyl
Drug: Tetracycline 125 MG — Antibiotic
  Other Names: Ambramicina
Drug: Bismuth Subcitrate — Antibiotic adjuvant
  Other Names: Denol
Drug: Rifabutin 150 MG — Antibiotic
  Other Names: Mycobutin
  Arms: Tailored therapy
Drug: Levofloxacin 500mg — Antibiotic
  Other Names: Levoxacin
  Arms: Tailored therapy

SUMMARY:
The aim of our study will be to assess in an open-label, multicenter, randomized controlled trial whether a tailored therapy guided by a non-invasive antibiotic susceptibility test on stool samples achieves higher Helicobacter eradication rates than an empiric antibiotic regimen. For this purpose, consecutive patients with dyspeptic symptoms, diagnosis of Helicobacter pylori infection and naïve to eradicating treatments will be allocated to either of the two intervention arms.

DETAILED DESCRIPTION:
Study design:

Eligible subjects will be defined by the positivity to at least 2 out of 4 tests for Helicobacter pylori infection diagnosis (i.e. histology, rapid urease test, urea breath test and serology). Stool samples and gastric biopsy specimens of eligible patients will be analyzed at enrollment, using real time-polymerase chain reaction (RT-PCR) to detect bacterial DNA mutations conferring resistance to amoxicillin, clarithromycin, tetracycline, metronidazole, and levofloxacin. Participants allocated to the tailored intervention arm will receive an antibiotic combination therapy according to the result of stool sample molecular analysis. Participants allocated to the empiric intervention arm will be treated by either a quadruple concomitant or bismuth-containing regimen, according to the 2017 European Helicobacter pylori management guidelines. In all participants, infection eradication will be evaluated 30 days after treatment end, using urea breath test. We will also assess the diagnostic accuracy of the RT-PCR on fecal samples in detecting bacterial antibiotic resistances, using the RT-PCR on gastric biopsy specimens as the reference standard.

ELIGIBILITY:
Inclusion Criteria:

* presence of dyspeptic symptoms, according to Rome IV criteria;
* Helicobacter pylori infection diagnosis by the positivity of at least 2 out of 4 diagnostic tests (i.e. histology, rapid urease test, urea breath test, and serology);
* naive to Helicobacter pylori treatment;
* written informed consent.

Exclusion Criteria:

* previous Helicobacter pylori treatment;
* diagnosis of gastric cancer or other diseases requiring surgery;
* contraindications to upper endoscopy;
* chronic diarrhea;
* known allergy to any drugs used in the intervention and control arm.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 362 (Estimated)
Dates: Start 2020-01-14 (Actual); Primary Completion 2021-02-14 (Estimated); Study Completion 2022-04-14 (Estimated)

PRIMARY OUTCOMES:
Eradication rate | 30 days
  Number of participants achieving Helicobacter pylori eradication

SECONDARY OUTCOMES:
Adverse events | 10 days
  Any adverse event occurring during the 10-day treatment
Participants' compliance | 10 days
  Number of assumed tablets divided by the total number of prescribed tablets
Treatment withdrawal | 10 days
  Withdrawal of any drug included in the prescribed regimen

OTHER OUTCOMES:
Diagnostic accuracy parameters | 30 days
  Sensitivity, specificity, positive predictive value, negative predictive value, positive and negative likelihood ratio, and accuracy of the RT-PCR on fecal samples for the detection of antibiotic resistances

CONTACTS AND LOCATIONS:
Overall Officials: Mariabeatrice Principi, Prof., Principal Investigator — University of Bari
Locations (1):
- Michele Barone, Bari, BA, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Malfertheiner P, Megraud F, O'Morain CA, Gisbert JP, Kuipers EJ, Axon AT, Bazzoli F, Gasbarrini A, Atherton J, Graham DY, Hunt R, Moayyedi P, Rokkas T, Rugge M, Selgrad M, Suerbaum S, Sugano K, El-Omar EM; European Helicobacter and Microbiota Study Group and Consensus panel. Management of Helicobacter pylori infection-the Maastricht V/Florence Consensus Report. Gut. 2017 Jan;66(1):6-30. doi: 10.1136/gutjnl-2016-312288. Epub 2016 Oct 5. PMID 27707777
- [Result] Iannone A, Giorgio F, Russo F, Riezzo G, Girardi B, Pricci M, Palmer SC, Barone M, Principi M, Strippoli GF, Di Leo A, Ierardi E. New fecal test for non-invasive Helicobacter pylori detection: A diagnostic accuracy study. World J Gastroenterol. 2018 Jul 21;24(27):3021-3029. doi: 10.3748/wjg.v24.i27.3021. PMID 30038469
- [Result] Giorgio F, Ierardi E, Sorrentino C, Principi M, Barone M, Losurdo G, Iannone A, Giangaspero A, Monno R, Di Leo A. Helicobacter pylori DNA isolation in the stool: an essential pre-requisite for bacterial noninvasive molecular analysis. Scand J Gastroenterol. 2016 Dec;51(12):1429-1432. doi: 10.1080/00365521.2016.1216592. Epub 2016 Aug 9. PMID 27687850
- [Result] Drossman DA. Functional Gastrointestinal Disorders: History, Pathophysiology, Clinical Features and Rome IV. Gastroenterology. 2016 Feb 19:S0016-5085(16)00223-7. doi: 10.1053/j.gastro.2016.02.032. Online ahead of print. PMID 27144617
- [Result] De Francesco V, Giorgio F, Hassan C, Manes G, Vannella L, Panella C, Ierardi E, Zullo A. Worldwide H. pylori antibiotic resistance: a systematic review. J Gastrointestin Liver Dis. 2010 Dec;19(4):409-14. PMID 21188333